CLINICAL TRIAL: NCT01821924
Title: Role of Stress CMR in Predicting Adverse Clinical Events in Patients With Known or Suspected Ischemic Heart Disease
Brief Title: Role of Stress CMR in Predicting Adverse Clinical Events in Patients With Known or Suspected IHD
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Raymond Y. Kwong, MD, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 2011P000643
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators plan to use retrospective data to assess heart function and structure abnormalities through the use of an approved vasodilating agent for stress cardiac MRI tests. The investigators are interested in how these MRI findings relate to long-term prognosis in people who are at risk for cardiac disease.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 21 years old
* No contraindications for cardiac MRI (by renal function or metallic hazards)

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients above the age of 21 who are clinically referred for stress cardiac MRI.
Sampling Method: Non-Probability Sample
Enrollment: 2347 (Actual)
Dates: Start 2012-01-30 (Actual); Primary Completion 2016-01-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
A composite outcome measure consisting of cardiovascular mortality and nonfatal MI after index CMR. | target follow up of at least 4 years
  "Myocardial infarction" will be defined as hospital admission for acute coronary syndrome (defined by positive serum troponin level with documented electrocardiographic changes, clinical syndrome, or need for percutaneous or surgical revascularization).

SECONDARY OUTCOMES:
A composite outcome measure consisting of cardiovascular mortality, nonfatal MI, hospitalization for unstable angina or congestive heart failure, and late unplanned coronary bypass surgery at at least 6 months after index CMR. | target follow up of at least 4 years
  "Heart failure hospitalization" will be defined as any hospitalization for signs and symptoms of volume overload or dyspnea requiring diuretic therapy regardless of LV ejection fraction.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Shah R, Heydari B, Coelho-Filho O, Murthy VL, Abbasi S, Feng JH, Pencina M, Neilan TG, Meadows JL, Francis S, Blankstein R, Steigner M, di Carli M, Jerosch-Herold M, Kwong RY. Stress cardiac magnetic resonance imaging provides effective cardiac risk reclassification in patients with known or suspected stable coronary artery disease. Circulation. 2013 Aug 6;128(6):605-14. doi: 10.1161/CIRCULATIONAHA.113.001430. Epub 2013 Jun 26. PMID 23804252